CLINICAL TRIAL: NCT03088904
Title: Genetic and Environmental Factors in the Response to Influenza Vaccination
Acronym: SLVP028
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 31050; 2U19AI057229-11 (NIH)
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Influenza; Healthy
Keywords: Inactivated influenza vaccine quadrivalent; Live, attenuated influenza vaccine quadrivalent; Monozygotic twins; Dizygotic twins; Adults; Adolescents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: MZ twins (IIV4) (Experimental): Group A: Up to 40 healthy monozygotic (MZ) individual twin volunteers, 12-49 years old, will be given inactivated influenza vaccine quadrivalent (IIV4) Fluzone® Quadrivalent vaccine. Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 6-8 and Day 28+7 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Fluzone® Quadrivalent vaccine
- Group B: DZ twins (IIV4) (Experimental): Group B: Up to 40 healthy dizygotic (DZ) individual twin volunteers, 12-49 years old, will be given inactivated influenza vaccine quadrivalent (IIV4) Fluzone® Quadrivalent vaccine. Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), and Day 6-8 and Day 28+ 7 (post-immunization). All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  Interventions: Biological: Fluzone® Quadrivalent vaccine
- Group C: MZ twins (IIV4 or LAIV4) (Experimental): Group C: Up to 40 healthy monozygotic (MZ) individual twin volunteers, 12-49 years old, will be randomized within the twin pair to receive either inactivated influenza vaccine quadrivalent (IIV4) Fluzone® Quadrivalent vaccine or live, attenuated influenza vaccine quadrivalent (LAIV4) FluMist® Quadrivalent. Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 6-8 and Day 28+7 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).
  This group was terminated in 2016 due to ACIP recommendations against the use of LAIV but may be reopened in 2018 pending LAIV4 availability.
  Interventions: Biological: FluMist® Quadrivalent; Biological: Fluzone® Quadrivalent vaccine

INTERVENTIONS:
Biological: FluMist® Quadrivalent — LAIV4 vaccine dosage is 0.2 mL. Vaccine will be administered as an intranasal spray. Each sprayer contains a single dose of FluMist® Quadrivalent; approximately one-half of the contents should be administered into each nostril. 0.1 mL (i.e., half of the dose from a single FluMist sprayer) is administered into each nostril while the recipient is in an upright position. Insert the tip of the sprayer just inside the nose and rapidly depress the plunger until the dose-divider clip stops the plunger. The dose divider clip is removed from the sprayer to administer the second half of the dose (0.1 mL) into the other nostril.
  Arms: Group C: MZ twins (IIV4 or LAIV4)
Biological: Fluzone® Quadrivalent vaccine — IIV4 vaccine will be administered as a 0.5 mL dose, with a sterile, disposable syringe and needle by IM injection into the deltoid muscle.

SUMMARY:
The purpose of the study is to investigate and compare the immune responses to influenza vaccination in monozygotic (identical) and dizygotic (fraternal) twins to determine the roles of genetics and environment in the response to flu vaccination.

DETAILED DESCRIPTION:
This is a phase 1 study of 120 healthy 12-49 year old adolescents and adult volunteers who are given licensed seasonal influenza vaccine. There are no exclusions for gender, ethnicity or race. The volunteers will be enrolled into one of 3 groups:

Group A: Up to 40 healthy monozygotic (MZ) twin volunteers, 12-49 years old, will be given inactivated influenza vaccine quadrivalent (IIV4). Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 6-8 and Day 28+ 7 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).

Group B: Up to 40 healthy dizygotic (DZ) twin volunteers, 12-49 years old, will be given inactivated influenza vaccine quadrivalent (IIV4). Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 6-8 and Day 28+7 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs).

Group C: Up to 40 healthy monozygotic (MZ) twin volunteers, 12-49 years old, will be randomized within the twin pair to receive either inactivated influenza vaccine quadrivalent (IIV4) or live, attenuated influenza vaccine quadrivalent (LAIV4). Each volunteer will complete a total of 3 visits: Day 0 (pre-immunization), Day 6-8 and Day 28+7 post-immunization. All visits will consist of drawing blood for study assays and monitoring for serious adverse events (SAEs). This group was terminated in 2016 due to ACIP recommendations against the use of LAIV but was reopened in 2018 with the availability of LAIV4.

Each twin is counted as a single participant. All reporting numbers reflect the number of participants, not the number of twin pairs.

ELIGIBILITY:
Inclusion Criteria

1. Otherwise healthy, 12-49 years old, identical (MZ) or fraternal (DZ) twins.
2. Willing to complete the informed consent process (including assent for minors 12-17 years of age, inclusive).
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history by review of inclusion/exclusion criteria and vital signs.

Exclusion Criteria

1. Prior off-study vaccination with the current year's seasonal influenza vaccine.
2. Allergy to egg or egg products, or to vaccine components, (including gentamicin, gelatin, arginine or MSG in LAIV)
3. Life-threatening reactions to previous influenza vaccinations.
4. Asthma (If yes, not eligible for Group C).
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination.
6. History of immunodeficiency (including HIV infection).
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Blood pressure >150 systolic or >95 diastolic at first study visit and the day of vaccination.
9. Hospitalization in the past year for congestive heart failure or emphysema.
10. Chronic Hepatitis B or C.
11. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible).
12. In close contact with anyone who has a severely weakened immune system and requires a protective environment (If yes, may be ineligible for Group C; exposure to such persons should be avoided for 7 days after receipt of LAIV).
13. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
14. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
15. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year.
16. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
17. For children or adolescents through 17 years of age, receiving aspirin therapy or aspirin-containing products (If yes, not eligible for Group C).
18. Receipt of blood or blood products within the past 6 months or planned used during the study.
19. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol.
20. Receipt of inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last study visit (~ 28 days after study vaccination).
21. Receipt of live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 28 days after study vaccination).
22. Need for allergy immunization (that cannot be postponed) during the study period.
23. Has taken an influenza antiviral medication within 48 hours prior to study vaccination (If yes, not eligible for Group C).
24. History of Guillain-Barré syndrome
25. Pregnant woman
26. Lactating woman (If yes, not eligible for Group C).
27. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
28. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned donation prior to completion of the last visit.
29. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 12 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition (HAI) titers in response to influenza vaccination. | Day 0 to Day 28
Interferon-gamma (IFN-γ) production by T cells | Day 0 to Day 28
IFN-γ production by Natural Killer (NK) cells. | Day 0 to Day 28

SECONDARY OUTCOMES:
Sequencing of T-cell receptor (TCR)ab and Immunoglobulin Genes | Day 0 to Day 28
  B and T cells will be sequenced for their antibody repertoires.
Natural Killer (NK) repertoire. | Day 0 to Day 28
  Mass cytometry will be used to assess the NK cell repertoire.

CONTACTS AND LOCATIONS:
Overall Officials: Mark M Davis, PhD, Principal Investigator — Stanford School of Medicine, Dept. of Microbiology and Immunology; Catherine Blish, MD, Principal Investigator — Stanford School of Medicine, Dept. of Medicine; William Robinson, MD, Principal Investigator — Stanford School of Medicine, Dept. of Medicine; Cornelia Dekker, MD, Principal Investigator — Stanford School of Medicine, Dept. of Pediatrics
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford-LPCH Vaccine Program Stanford University School of Medicine — http://vaccines.stanford.edu/